CLINICAL TRIAL: NCT06645184
Title: Effects of Adding Appetite Stimulants to a Fibre Containing High-Protein ONS on Appetite-Related Outcomes in Older Adults
Brief Title: Adding Appetite Stimulants to an ONS in Older Adults
Acronym: APPOLO II
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nutricia Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: 24REX0063741
Record Dates: First submitted 2024-10-08; First posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Malnutrition
MeSH Terms: conditions — Malnutrition | interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Participating subjects are blinded and will not know which of the 4 study products they will consume
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- ONS with fibre with added nutrients (Other)
  Interventions: Dietary Supplement: Oral nutritional supplement
- ONS without fiber with added nutrients (Other)
  Interventions: Dietary Supplement: Oral nutritional supplement
- ONS with fibre without added nutrients (Other)
  Interventions: Dietary Supplement: Oral nutritional supplement
- ONS without fibre without added nutrients (Other)
  Interventions: Dietary Supplement: Oral nutritional supplement

INTERVENTIONS:
Dietary Supplement: Oral nutritional supplement — During 4 test days, 1 bottle (125ML) of High protein ONS with or without fibre and with or without the added nutrients will be consumed by the subjects. During each test day, the subjects will complete questionnaires related to appetite and liking of the product from baseline (-5 minutes of start consumption of study product) until 120 minutes after start consumption of study product.

SUMMARY:
Study to determine whether adding specific nutrients to a high-protein oral nutritional support (ONS), with and without fibre can reduce the feeling of satiety and may increase appetite in adults older than 65 years. This contributes to research into a new type of nutritional nutrition for people with disease related malnutrition (DRM)

ELIGIBILITY:
Inclusion Criteria:

1. 65 years of age or older
2. Able to consume high energy and/or high protein ONS at discretion of the Investigator
3. Written informed consent
4. Willing and able to refrain from smoking during the visits
5. Able to speak and read in Dutch to communicate with the site staff and comply with the instructions and requirements of the study.

Exclusion Criteria:

1. Any known condition that interferes with the gastric emptying (e.g., gastroparesis, gastric stoma, hypothyroidism, hyperthyroidism, multiple sclerosis, Parkinson disease).
2. Any known metabolic condition that interferes with the breakdown of amino acids (e.g. arginase deficiency, urea cycle disorder)
3. Known history of gastric surgery e.g. (partial) gastrectomy or any other procedure for stomach volume reduction, including gastric banding, gastric balloon.
4. Any known chronic/continuous use, and/or within 24-48h before the visit, of medication that strongly affects with gastric emptying or gastric acid secretion (e.g., metoclopramide, opioid analgesics, calcium channel blockers, Beta-Adrenergic Receptor Agonists, H2 receptor antagonists, proton pump inhibitors; tricyclic antidepressants such as amitriptyline, imipramine, systemic steroids)
5. Known active cancer treatment 4 weeks prior the study start
6. Body Mass Index >= 30.0 kg/m²
7. Presence of Diabetes Mellitus (self-reported or the use of Diabetes medication: i.e., insulin, biguanides, DPP-4 inhibitors, GLP-1 receptor agonists)
8. Investigator's uncertainty about the willingness or ability of the subject to comply with the protocol requirements, for example due to the presence of a psychiatric disorder (e.g. major depression, psychoses), dementia or Alzheimer's disease
9. Known renal dysfunction with protein restriction diet
10. Known allergy to cow's milk protein
11. Known allergy to soy
12. Known galactosaemia
13. Known lactose intolerance
14. Excessive alcohol consumption (use of > 14 units per week for women or > 21 units per week for men, on average during the past 6 months).
15. Drug abuse based on investigator's judgement.
16. Any contraindication to oral feeding per se being: any degree of dysphagia, gastrointestinal failure or suppressed gastrointestinal function, complete intestinal obstruction and major intra-abdominal sepsis.
17. Enrolment in any other studies involving investigational or marketed products concomitantly or within two weeks prior to baseline
18. Employees, family members or other relatives of employees of the participating centre or of Danone Global Research & Innovation Center.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
composite satiety score (CSS) | 120 minutes
  The main outcome parameter in this study is the composite satiety score (CSS), measured from baseline (-5 minutes) until 120 minutes after starting the consumption of the study product.

SECONDARY OUTCOMES:
Satiety after 120 min | more than 120 minutes
  Satiety, fullness, hunger, prospective food consumption measured from baseline until 120 minutes after starting the consumption of the study product measured with composite satiety score questionnaire
Volume consumed | 120 minutes
  Adherence to use of the study product, defined as volume consumed within 10 minutes relative to 1 serving [%]

IPD SHARING:
Plan to Share IPD: No